CLINICAL TRIAL: NCT06099145
Title: Clinical and Medico-economic Study to Validate the Performance of a Digital and Personalized Solution (HEPHAÏ) to Support the Use of Inhaled Treatments for Asthma and COPD
Brief Title: Clinical and Medico-economic Validation of the HEPHAI Solution.
Acronym: VAL-HEPHAI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hephai (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KM00385
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Asthma COPD

STUDY DESIGN:
Intervention Model Description: This is an interventional, multicenter, randomized, controlled clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patient who received inhaled treatment with Innovair® or Trimbow® as a part standard care for 6 months
- Hephai (Experimental): Patient using the Hephaï medical device as a tool who received inhaled treatment with Innovair® or Trimbow® as a part standard care for 6 months
  Interventions: Device: Hephaï

INTERVENTIONS:
Device: Hephaï — Used of the HEPHAI medical device as a tool to improve the delivery of inhaled treatments for asthma and COPD
  Arms: Hephai

SUMMARY:
In a context where the use of inhalation devices for respiratory medications is associated with a high frequency of critical errors, our primary hypothesis is that the use of the HEPHAÏ solution reduces this frequency compared to standard care.

The objective of this clinical study is to evaluate the performance of the HEPHAÏ solution as a tool for improving the administration of inhaled treatments in patients undergoing pulmonary care for asthma and/or COPD, who are receiving treatment with Innovair® or Trimbow®. These two inhalers were chosen for reasons of feasibility and compatibility with the version of the HEPHAÏ software provided as part of the clinical investigation

DETAILED DESCRIPTION:
The proper use of inhalation devices is crucial to relieving asthma and COPD symptoms and preventing exacerbations of these diseases. The improper use of these devices is currently considered a major problem. HEPHAI (Class I Medical Device) is a versatile application based on artificial intelligence (AI), allowing to recognize the appropriate use of an inhalation device by analyzing (without any sensors either on the patient or on the inhaler), the sequence of movements and sounds necessary for error-free intake. The HEPHAI application allows the patient to film themselves directly when using their inhaler, to interrogate in real time an AI based on behavior recognition (movements and sounds), to give the patient an immediate result, and to set up a corrective process if the intake has not been properly carried out.

HEPHAÏ is thus a companion tool to the inhaler prescribed by the doctor, which allows the patient to benefit from assistance in the use of his or her personalized inhaler at home.

Among patients using an inhalation device for their treatment, 30% to 40% make errors of use that are considered "critical", i.e. making the treatment ineffective or drastically reducing its effectiveness. Beyond its clinical impact (persistence of symptoms, decreased adherence, increased risk of exacerbation), the economic cost of this inadequate use is estimated at nearly one billion euros per year in France, with a major weight of hospitalizations for exacerbations.

In this contaxt, the objective of the present study is to evaluate the performance of the HEPHAÏ solution as a tool for improving the administration of inhaled treatments in patients undergoing pulmonary care for asthma and/or COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age
* Patient followed in pulmonology for Asthma and/or COPD with implementation and/or follow-up of treatment with Innovair® or Trimbow®,
* Patient affiliated to a Social Security scheme,
* Patient with a hardware support allowing the operation of HEPHAÏ: smartphone, tablet, desktop or laptop computer with graphical interface, video, sound and a high-speed connection at the place of use.

Exclusion Criteria:

* Patient previously enrolled in another interventional clinical study,
* Adult patients who are subject to a legal protection measure (guardianship, judicial safeguard, psychiatric care or deprived of liberty by judicial or administrative decision),
* Patient with at least one sensory, visual or tactile impairment, preventing the correct use of a smartphone, tablet and/or computer or preventing the correct performance of the exercise safely,
* Patient with a cognitive impairment, severely limiting their ability to concentrate and thus preventing the correct use of a smartphone, tablet and/or computer,
* Patient cared for by a specialized team of education, therapeutic for his asthma or COPD follow-up (e.g. asthma school, asthma referent IDE),
* Patient who does not understand French,
* Patient with an inhalation chamber prescription associated with their inhalation device prescription.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Critical Errors at week 12 | Baseline and week 12
  Assessment of the proportion of critical errors during inhaler use, from baseline to 3 months after initiation of the intervention.
  A critical error is defined as an error during use of the device that would compromise access of the inhaled medication to the respiratory tract, The methodology used to assess critical errors consists in comparing the results of the investigating physician's observation of use with a reference checklist developed on the basis of official recommendations for use.

SECONDARY OUTCOMES:
Proportion of Critical Errors at week 24 | Baseline to week 24
  Assessment of the proportion of critical errors during inhaler use, from baseline to 6 months after initiation of the intervention.
  A critical error is defined as an error during use of the device that would compromise access of the inhaled medication to the respiratory tract, The methodology used to assess critical errors consists in comparing the results of the investigating physician's observation of use with a reference checklist developed on the basis of official recommendations for use.
Quality of Life Assessment (Saint-Georges' Hospital Questionnaire) | Baseline to week 24
  Assessment of quality of life using the Saint-Georges' Hospital questionnaire (French version) at each time, with a specific focus on the evolution from baseline to week 24
Quality of Life Assessment (EQ5D5L Questionnaire) | Baseline to week 24
  Assessment of quality of life using the EQ5D5L questionnaire at each time, with a specific focus on the evolution from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Capucine.morelot@aphp.fr, Prof., Principal Investigator — Department of Pneumonology, Pitié-Salpêtrière Hospital,
Locations (5):
- France (5):
  - CHU de Dijon, Dijon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Pitié-Salpêtrière Hospital, Paris
  - Hôpital COCHIN, Paris
  - Hôpital BICHAT, Paris